CLINICAL TRIAL: NCT01588327
Title: A Prospective Pharmacodynamic Study of Dabigatran Using Peak and Trough Coagulation Test Results in Patients on Therapeutic Doses of Dabigatran
Brief Title: A Prospective Pharmacodynamic Study of Dabigatran
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 11-1693
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Blood Coagulation Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental: Patient taking FDA approved dose of dabigatran
- Control group: Person not taking any form of anticoagulation.

SUMMARY:
The ability to explain bleeding or clotting complications in patients treated with dabigatran remains challenging. In addition, there is limited data on how coagulation tests perform in patients treated with therapeutic doses of dabigatran. Predicted responses of coagulation tests to therapeutic doses of dabigatran may be helpful in better understanding abnormal responses to dabigatran. The purpose of the study is to define a therapeutic reference range for peak and trough coagulation tests in patients taking FDA approved doses of dabigatran and to determine which tests may be most clinically useful for monitoring dabigatran.

ELIGIBILITY:
Inclusion Criteria:

• Medication therapy with dabigatran 75 mg twice daily or 150 mg twice daily for a minimum of 3 days

Exclusion Criteria:

* CrCl < 15 ml/min
* Non-FDA approved dose based on calculated CrCl with most recent SCr
* Age < 18 years
* Inability to communicate in the English language
* Decisionally-impaired individuals
* Incarcerated
* Pregnant/Lactating (Pregnancy category: C, unevaluated effects in lactation)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients taking FDA-approved doses of dabigatran and control subjects not taking an anticoagulant or antiplatelet were eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Hawes, PharmD, Principal Investigator — University of North Carolina, Chapel Hill

REFERENCES:
- [Derived] Hawes EM, Deal AM, Funk-Adcock D, Gosselin R, Jeanneret C, Cook AM, Taylor JM, Whinna HC, Winkler AM, Moll S. Performance of coagulation tests in patients on therapeutic doses of dabigatran: a cross-sectional pharmacodynamic study based on peak and trough plasma levels. J Thromb Haemost. 2013 Aug;11(8):1493-502. doi: 10.1111/jth.12308. PMID 23718677